CLINICAL TRIAL: NCT01833260
Title: Influence of a Distractive Auditory Stimulus on the Rate of Exertion During Pulmonary Rehabilitation Sessions
Brief Title: Music and Perceived Rate of Exertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Doctor in Physiotherapy, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Music
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With music (Experimental): Pulmonary rehabilitation with music in the room
  Interventions: Behavioral: Music
- Without music (No Intervention)

INTERVENTIONS:
Behavioral: Music
  Arms: With music

SUMMARY:
The aim of this study was to evaluate the effect of listening to ambient music on the perceived exertion rate during pulmonary rehabilitation for chronic obstructive pulmonary disease patients.

ELIGIBILITY:
Inclusion Criteria:

* participate in the program for at least one month after the initial medical investigation, be free of exacerbations for 1 month and have maintained exactly the same program session for both evaluated sessions

Exclusion Criteria:

* participate to only session of one condition

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Rate of exertion | After 1 hour

SECONDARY OUTCOMES:
Dyspnea | After 1 hour
  Using a visual analogue scale
Hospital Anxiety Depression Scale | After 1 hour
  The score of anxiety and depression will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Reychler G, Mottart F, Boland M, Wasterlain E, Pieters T, Caty G, Liistro G. Influence of ambient music on perceived exertion during a pulmonary rehabilitation session: a randomized crossover study. Respir Care. 2015 May;60(5):711-7. doi: 10.4187/respcare.03671. Epub 2015 Jan 13. PMID 25587172